CLINICAL TRIAL: NCT07140159
Title: Recurrent Neural Networks for Windlass Mechanism Subphase Recognition and Anthropometric Angles Monitoring
Brief Title: Biomechanical Analysis of Gait
Status: Completed | Type: Observational
Sponsor: Universidad Politécnica de Baja California (Other)
Responsible Party: Principal Investigator, Gabriel Trujillo-Hernández, Research-Professor, Universidad Politécnica de Baja California
Other Study IDs: Approval Number 02/25
Record Dates: First submitted 2025-08-06; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Biomechanical Assessment of the Foot During Gait

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal gait group

SUMMARY:
This study measures the medial longitudinal arch angle and the metatarsophalangeal angle during the gait cycle in 35 healthy participants using speed cameras and reflective markers placed on anthropometric points.

DETAILED DESCRIPTION:
The medial longitudinal arch angle comprises the calcaneus, navicular tuberosity, and the head of the 1st metatarsal, while the metatarsophalangeal angle comprises the head of the 1st metatarsal and the proximal interphalangeal joint of the toe. These measurements provide valuable information on the stress of the plantar fascia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Aged between 18 and 43 years
* Foot sizes ranging from US 5 to 12
* Body weights between 53 to 125 kg
* Heights from 1.49 to 1.90 m
* BMI ranging from 21.8 to 39.9 kg/m².

Exclusion Criteria:

* Pes planus (flatfoot)
* Pes cavus (high-arched foot)
* Valgus rearfoot
* Varus rearfoot
* Foot deformities

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers aged 18 to 43 years, with no history of foot deformities.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Metatarsophalangeal Joint Angle | Baseline
  This angle comprises the supplementary angle formed by the first metatarsal head, posterior calcaneus, and proximal interphalangeal. The angle is measured using a marker-based motion capture system with blue markers placed on these points and recorded with cameras operating at 60 frames per second. A centroid-based landmark detection algorithm determines the centroid coordinates and applies trigonometric functions to each frame to calculate the angle in degrees with a precision of two decimal places.
Medial Longitudinal Arch Angle | Baseline
  This angle is defined by the anthropometric landmarks of the calcaneus, the navicular tuberosity, and the head of the first metatarsal. The angle is measured using a marker-based motion capture system with blue markers placed on these points and recorded with cameras operating at 60 frames per second. A centroid-based landmark detection algorithm determines the centroid coordinates and applies trigonometric functions to each frame to calculate the angle in degrees with a precision of two decimal places.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad politécnica de baja california, Mexicali, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.youtube.com/watch?v=dLADQdmE2nk